CLINICAL TRIAL: NCT03195075
Title: Endoscopic Ultrasonography-Guided Biliary Drainage Versus Percutaneous Trans-hepatic Biliary Drainage for Malignant Biliary Obstruction After Failed Endoscopic Retrograde Cholangio-pancreaticography
Brief Title: Endoscopic Ultrasonography Guided Biliary Drainage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelhamed Mohamed, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUS
Record Dates: First submitted 2017-06-04; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Malignant Hepatobiliary Neoplasm

STUDY DESIGN:
Intervention Model Description: This study will include 40 consecutive jaundiced patients with distal malignant biliary obstruction after failed endoscopic retrograde cholangio-pancreaticography. Twenty patients with failed endoscopic retrograde cholangio-pancreaticography will be subjected to endoscopic ultrasonography-guided biliary drainage will be performed by single endoscopist and another 20 patients with failed endoscopic retrograde cholangio-pancreaticography for percutaneous trans-hepatic biliary drainage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): 20 Patients with malignant biliary obstruction after failed endoscopic retrograde cholangio-pancreaticography will be subjected to endoscopic ultrasonography guided biliary drainage
  Interventions: Procedure: Endoscopic ultrasonography guided biliary drainage
- Group 2 (Active Comparator): 20 Patients with malignant biliary obstruction after failed endoscopic retrograde cholangio-pancreaticography will be subjected to percutaneous trans-hepatic biliary drainage.
  Interventions: Procedure: Percutaneous trans-hepatic biliary drainage

INTERVENTIONS:
Procedure: Endoscopic ultrasonography guided biliary drainage — Endoscopic ultrasonography guided biliary drainage includes rendezvous techniques, endoscopic ultrasonography guided choledochoduodenostomy, and endoscopic ultrasonography-guided hepatogastrostomy using self-expandable metal stent will be done for group 1
  Arms: Group 1
Procedure: Percutaneous trans-hepatic biliary drainage — Percutaneous trans-hepatic biliary drainage in interventional radiology department using self-expandable metal stent will be done for group 2
  Arms: Group 2

SUMMARY:
Endoscopic ultrasonography is a widely accepted modality for the diagnosis of gastrointestinal and pancreatic-biliary diseases.

Endoscopic ultrasonography-guided biliary drainage has attracted attention as an alternative procedure to percutaneous trans-hepatic biliary drainage, with a technical success between 75%-100% and with low complication rate. Other important advantage of endoscopic ultrasonography-guided biliary drainage compared with external percutaneous trans-hepatic biliary drainage is better quality of life due to the internal placement of the stent.

DETAILED DESCRIPTION:
If endoscopic retrograde cholangio-pancreaticography fails to achieve biliary drainage, more invasive options are usually considered. These include percutaneous trans-hepatic biliary drainage and surgical intervention but they have been associated with a higher risk of complications and prolonged hospital stay.

Some disadvantages with the percutaneous approach include the need to traverse the liver, a decreased quality of life due to the presence of external drainage and a significant morbidity and mortality, 7% and 5% respectively.

The external drainage of percutaneous trans-hepatic biliary drainage may add to the patient's burden owing to the cosmetic problem, skin inflammation or pain, or bile leakage, compromising the quality of life. From this point, the internal drainage of endoscopic ultrasonography-guided biliary drainage eliminates several issues.

Endoscopic ultrasonography-guided biliary drainage using a metal stent, particularly a lumen-apposing metal stent, can also be performed in patients with a large amount of ascites, which is often contraindicated in percutaneous trans-hepatic biliary drainage. Endoscopic ultrasonography-guided biliary drainage performed in the same session of the failed endoscopic retrograde cholangio-pancreaticography, in the same room and under the same sedation.

On the other hand, the endoscopic ultrasonography-guided biliary drainage, has major limitation due to fewer cases reported till date and lack of long term data. Because of, the technical difficulty encountered during re-intervention and problem of stent migration, the expertise needed for such procedure is a major limitation of the techniques.

Furthermore, comparative studies of endoscopic ultrasonography-guided biliary drainage versus percutaneous trans-hepatic biliary drainage are required to select the optimal candidates and to best evaluate the technical and treatment outcomes also in terms of quality of life and costs. Recently, Endoscopic ultrasonography-guided biliary drainage has been introduced as an alternative for patients who had failed endoscopic retrograde cholangio-pancreaticography.

Indications for endoscopic ultrasonography-guided biliary drainage:

1. Failed conventional endoscopic retrograde cholangio-pancreaticography.
2. Altered anatomy
3. Tumor preventing access into the biliary tree
4. Prior surgical procedure
5. Biliary sphincter stenosis
6. Contra-indication to percutaneous access

ELIGIBILITY:
Inclusion Criteria:

1. Presence of un-resectable malignant distal biliary obstruction.
2. Failed conventional endoscopic retrograde cholangio-pancreaticography and inaccessible papilla because of accompanying duodenal obstruction, peri-ampullary tumor infiltration, ampulla stenosis, or surgically altered anatomy (Billroth II operation, Roux-an-Y operation).
3. Histological or cytological diagnosis of malignancy
4. No serious or uncontrolled medical illness

Exclusion Criteria:

1. Patient age of less than 18 years
2. Uncorrectable coagulopathy
3. History of allergy to radio-contrast agents
4. Refusal to participate in this study
5. Severs co-existed cardiopulmonary and /or renal disease
6. Low platelet count (50000/μL)
7. Patients with disturbed conscious level

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Laboratory evaluation of efficacy of endoscopic ultrasonography and percutaneous trans-hepatic biliary drainage in malignant biliary obstruction. | Liver function test before the procedure and follow up changes after one week from procedures.
  Evaluation of serum bilirubin and alkaline phosphatase by liver function test before and after the procedures
Radiological evaluation of efficacy of endoscopic ultrasonography and percutaneous trans-hepatic biliary drainage in malignant biliary obstruction | Biliary dilation before the procedures and follow up changes after one week from procedures.
  Evaluation of biliary dilation by abdominal ultrasonography before and after the procedures,

SECONDARY OUTCOMES:
Evaluation of post-procedural complications | Within six months from procedure.
  Evaluation of biliary leakage by ultrasound, hemorrhage by hemoglobin level, perforation and stent potency.

REFERENCES:
- [Background] Ferrucci JT Jr, Mueller PR, Harbin WP. Percutaneous transhepatic biliary drainage: technique, results, and applications. Radiology. 1980 Apr;135(1):1-13. doi: 10.1148/radiology.135.1.7360943.
- [Background] Vilmann P, Jacobsen GK, Henriksen FW, Hancke S. Endoscopic ultrasonography with guided fine needle aspiration biopsy in pancreatic disease. Gastrointest Endosc. 1992 Mar-Apr;38(2):172-3. doi: 10.1016/s0016-5107(92)70385-x. No abstract available. PMID 1568614
- [Background] Hanada K, Iiboshi T, Ishii Y. Endoscopic ultrasound-guided choledochoduodenostomy for palliative biliary drainage in cases with inoperable pancreas head carcinoma. Dig Endosc. 2009 Jul;21 Suppl 1:S75-8. doi: 10.1111/j.1443-1661.2009.00855.x. PMID 19691742
- [Background] Collins D, Penman I, Mishra G, Draganov P. EUS-guided celiac block and neurolysis. Endoscopy. 2006 Sep;38(9):935-9. doi: 10.1055/s-2006-944734. PMID 16981114
- [Background] van der Gaag NA, Rauws EA, van Eijck CH, Bruno MJ, van der Harst E, Kubben FJ, Gerritsen JJ, Greve JW, Gerhards MF, de Hingh IH, Klinkenbijl JH, Nio CY, de Castro SM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for cancer of the head of the pancreas. N Engl J Med. 2010 Jan 14;362(2):129-37. doi: 10.1056/NEJMoa0903230. PMID 20071702
- [Background] Puspok A, Lomoschitz F, Dejaco C, Hejna M, Sautner T, Gangl A. Endoscopic ultrasound guided therapy of benign and malignant biliary obstruction: a case series. Am J Gastroenterol. 2005 Aug;100(8):1743-7. doi: 10.1111/j.1572-0241.2005.41806.x. PMID 16086710
- [Background] Shami VM, Kahaleh M. Endoscopic ultrasonography (EUS)-guided access and therapy of pancreatico-biliary disorders: EUS-guided cholangio and pancreatic drainage. Gastrointest Endosc Clin N Am. 2007 Jul;17(3):581-93, vii-viii. doi: 10.1016/j.giec.2007.05.015. PMID 17640584
- [Background] Fabbri C, Luigiano C, Lisotti A, Cennamo V, Virgilio C, Caletti G, Fusaroli P. Endoscopic ultrasound-guided treatments: are we getting evidence based--a systematic review. World J Gastroenterol. 2014 Jul 14;20(26):8424-48. doi: 10.3748/wjg.v20.i26.8424. PMID 25024600
- [Background] Mallery S, Matlock J, Freeman ML. EUS-guided rendezvous drainage of obstructed biliary and pancreatic ducts: Report of 6 cases. Gastrointest Endosc. 2004 Jan;59(1):100-7. doi: 10.1016/s0016-5107(03)02300-9. PMID 14722561
- [Background] Kim YS, Gupta K, Mallery S, Li R, Kinney T, Freeman ML. Endoscopic ultrasound rendezvous for bile duct access using a transduodenal approach: cumulative experience at a single center. A case series. Endoscopy. 2010 Jun;42(6):496-502. doi: 10.1055/s-0029-1244082. Epub 2010 Apr 23. PMID 20419625
- [Background] Artifon EL, Ferreira FC, Otoch JP, Rasslan S, Itoi T, Perez-Miranda M. EUS-guided biliary drainage: a review article. JOP. 2012 Jan 10;13(1):7-17. PMID 22233941
- [Background] Artifon EL, Okawa L, Takada J, Gupta K, Moura EG, Sakai P. EUS-guided choledochoantrostomy: an alternative for biliary drainage in unresectable pancreatic cancer with duodenal invasion. Gastrointest Endosc. 2011 Jun;73(6):1317-20. doi: 10.1016/j.gie.2010.10.041. Epub 2010 Dec 31. No abstract available. PMID 21195404
- [Background] Burmester E, Niehaus J, Leineweber T, Huetteroth T. EUS-cholangio-drainage of the bile duct: report of 4 cases. Gastrointest Endosc. 2003 Feb;57(2):246-51. doi: 10.1067/mge.2003.85. PMID 12556796